CLINICAL TRIAL: NCT07105696
Title: The Effectiveness of the Web-Based CORE on Nursing Students' Health Diagnosis Skills: A Randomized Controlled Trial
Brief Title: The Effectiveness of the Web-Based CORE on Nursing Students' Health Diagnosis Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Gamze Bolattürk, Doctor Research Assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CORE-RCT-2025
Record Dates: First submitted 2025-07-13; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Health Diagnosis Skills; CORE; Nursing Students; Clinical Oriented Reasoning Exam

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the randomization process, those who meet the criteria for inclusion in the sample and accept to participate in the study do not know that they will be included in the intervention group or the control group, so it will be single-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based CORE (Experimental): The intervention planned for the study is a web-based digital CORE method. Students in the intervention group taking the Health Diagnosis course will be administered a web-based digital CORE to assess the cardiovascular, respiratory, musculoskeletal, and gastrointestinal systems.
  Interventions: Other: Web-Based CORE
- Control Group (No Intervention): Control group students will be asked the same multiple-choice questions in a digital environment, assessing the cardiovascular, respiratory, musculoskeletal, and gastrointestinal systems.

INTERVENTIONS:
Other: Web-Based CORE — The intervention planned for the study is a web-based digital CORE method. Students in the intervention group taking the Health Diagnosis course will be administered a web-based digital CORE to assess the cardiovascular, respiratory, musculoskeletal, and gastrointestinal systems.
  Students in the experimental group will be administered the web-based digital CORE exam. Students in the control group will be asked the same multiple-choice questions in a digital environment. Two weeks later, students in the experimental and control groups will be administered another exam. Differences in achievement scores between the two groups will be evaluated.
  Arms: Web-Based CORE

SUMMARY:
Health diagnosis is an essential part of the professional nursing role and the holistic nursing approach. The goal of the health diagnosis process is to establish a baseline database for the care plan, encompassing the patient's health status, risk factors related to their current health status, and health education needs. This process involves obtaining the patient's health history, conducting a physical examination, collecting other relevant data from the patient's health records, and recording the data identified. Collecting and analyzing information about the patient's health status begins with diagnosis. Diagnosis is the comprehensive and systematic process of collecting data to obtain information about the patient's current and past health status and to identify coping strategies used in cases of health deviations. Diagnosis enables the creation of a comprehensive database of the patient's health status. Therefore, one of the most important stages of the diagnostic process is the physical examination. The purpose of the physical examination is to collect detailed, objective data regarding the patient's physiological state. Physical examination is the ability to interpret what is seen, heard, and felt regarding the patient's condition. Inspection, palpation, auscultation, and percussion methods allow for the validation of data obtained through the nursing history and the acquisition of new data. Appropriate, accurate, and timely health diagnosis is the cornerstone of maintaining patient safety. Furthermore, because health diagnosis and physical examination require a comprehensive assessment of all body systems, they also facilitate improved communication and collaboration among nurses, patients, and other healthcare team members. Therefore, health diagnosis is an important component of nursing education.

Health diagnosis is a clinical problem. Decision-making is one of the most important skills required to solve a clinical problem. In nursing education, curricula need to be developed to develop clinical thinking and problem-solving skills in students.

There is often no single right or wrong in the relationship between the patient and the nurse. In such cases, the Clinically Oriented Reasoning Exam (CORE) is used to teach cause-effect relationships. CORE develops reasoning skills in decision-making. The classic CORE application is conducted in a laboratory setting. Each table in the laboratory is considered a station, and for each station, a clinical case is prepared in a format the student can understand. Information about the case is recorded on the front and back of the cards. The student is asked to answer, and depending on the correct step level, the student is given a negative or positive score. When the student turns the card over, they receive feedback on the question. The first student and the observer go to the first station, where the student reads the case and turns over as many cards as they want. Each card turned over is recorded. When a station is completed, the cards are rearranged to their original positions, and the student and observer move on to the next station. Another student returns with their observer to the previous station. Completion of all stations signifies completion of the exam.

Conducting the traditional CORE is time-consuming and difficult. To eliminate the disadvantages of CORE and make the exam more effective, a web-based application method will be used. This will facilitate the assessment phase. The research was planned as a randomized controlled experimental study. The research question for this study was to determine the effectiveness of the digital CORE application on health diagnostic skills. Additionally, the relationships between the digital CORE application and demographic variables will be examined. The findings will be discussed with the contribution of literature, and recommendations for further research will be presented. The findings will provide insights into the variables associated with the digital CORE application, skill effectiveness, and achievement.

ELIGIBILITY:
Inclusion Criteria:

* first-time enrollment in a health diagnosis course
* volunteering to participate in the study

Exclusion Criteria:

* not attending class and being absent
* not wanting to participate in research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical reasoning performance measured by the web-based Clinical Oriented Reasoning Exam (CORE) [Score range: 0-100; higher scores indicate better performance] | Week 4 (immediately after completion of the four-week module covering gastrointestinal, respiratory, cardiovascular, and musculoskeletal system assessments)
  The CORE is a standardized web-based test that evaluates students' clinical reasoning skills through case-based scenarios. It is administered at the conclusion of the four-week educational program, and results will be aggregated and reported as mean ± standard deviation (SD).

SECONDARY OUTCOMES:
Knowledge retention measured by the follow-up recall quiz [Score range: 0-100; higher scores indicate better retention] | Week 6 (two weeks after completion of the web-based Clinical Oriented Reasoning Exam [CORE])
  A standardized online recall quiz is administered two weeks after the CORE to assess retention of clinical reasoning knowledge gained during the four-week module. Quiz scores will be reported as mean ± standard deviation (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No